CLINICAL TRIAL: NCT05006001
Title: Evaluation of Colchicine and Nonsteroidal Anti-inflammatory Drug Combination Therapy and Renal Function in Gout Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: En Chu Kong Hospital (Other)
Responsible Party: Principal Investigator, Ya-Ling Huang, Principal Investigator, En Chu Kong Hospital
Other Study IDs: EnChuKongH
Record Dates: First submitted 2021-05-27; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Renal Impairment; Gout; Colchicine Adverse Reaction; Nonsteroidals (NSAIDs)Toxicity
Keywords: Acute kidney injury; Renal impairment; Nonsteroidal antiinflammatory drug; Drug-drug interaction
MeSH Terms: conditions — Renal Insufficiency; Gout; Acute Kidney Injury | interventions — Colchicine; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Case: Cases were defined as patients with an event of renal impairment during follow-up, such as acute kidney injury.
  Interventions: Drug: Colchicine and NSAID
- Control: Cases were defined as patients without an event of renal impairment during follow-up, such as acute kidney injury.
  Interventions: Drug: Colchicine and NSAID
- Exposure: Exposure was defined as patients with colchicine and NSAIDs combination therapy.
- Non-Exposure: Non-Exposure was defined as patients with other gout therapy.

INTERVENTIONS:
Drug: Colchicine and NSAID — Colchicine and nonsteroidal anti-inflammatory drug combination therapy
  Groups: Case; Control

SUMMARY:
Our findings are expected to provide real-world evidence of the renal-adverse effects of colchicine and NSAIDs combination therapy in patients with gout, which will guide healthcare professions in optimizing gout treatment regimens and evaluating risks of renal impairment.

DETAILED DESCRIPTION:
Background: Gout is a common prevalent disease, which causes a low quality of life and poses a significant health burden nationally and internationally. Colchicine and Nonsteroidal anti-inflammatory drug (NSAID) are the mainstay treatment of gout. Concurrent use of colchicine and NSAIDs are more than half in all prescriptions of the gout patients. Both colchicine and NSAIDs may cause renal impairment. However, the empirical evidence of renal impairment of colchicine and NSAIDs combination therapy is limited and even absent.

Objectives: This proposal will assess the association between colchicine and NSAIDs combination therapy and acute kidney injury. The investigators further evaluate the relationships of duration-response, recency-response, and dose-response.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a gout diagnosis
* Initially receiving at least one anti-gout drug

Exclusion Criteria:

* <1 year of continuous health insurance enrollment
* Colchicine and NSAID use before the cohort entry date
* Patients with hemodialysis or peritoneal dialysis before the cohort entry date
* Patients with acute kidney injury before the cohort entry date

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with gout and initiating anti-gout drug
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | Through study completion, an average of 1 year
  Number of participants with a diagnosis of acute kidney injury

SECONDARY OUTCOMES:
All cause mortality | Through study completion, an average of 1 year
  Number of participants with a death record
Hemodialysis or peritoneal dialysis | Through study completion, an average of 1 year
  Number of participants with a dialysis record

IPD SHARING:
Plan to Share IPD: Undecided